CLINICAL TRIAL: NCT04484090
Title: Safety and Efficacy of Ohhmed Treatments for the Improvement of Erectile Dysfunction - A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHH-MED Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHH-FE-0.1
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vertica (Experimental): Treatment with Vertica RF device for improving erectile function for men with erectile dysfunction
  Interventions: Device: Vertica RF device

INTERVENTIONS:
Device: Vertica RF device — The treatment provided by the Vertica device is indicated for improving the erectile function in men with erectile dysfunction

SUMMARY:
Erectile dysfunction, the persistent inability to achieve or maintain an erection sufficient for satisfactory sexual performance, is estimated to affect up to 30 million men in the United States. The disorder is age-associated. The available treatments include oral therapy, vacuum-constriction devices; shockwave therapy, intracavernosal injections of vasoactive agents, including alprostadil (prostaglandin E1, transurethral delivery of alprostadil, Implantation of penile prostheses.

The OhhMed Company has developed the Vertica device that provides treatments for improvement of erectile function in patients with erectile dysfunction. This study assess the safety, efficacy, ease of use, and satisfaction of the Vertica device by men with mild to moderate erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* IIEF-EF score of 11-24 with or without the use of medication (PDE5 inhibitors).
* Erectile dysfunction for at least 3- months
* Steady relationship for at least 3-months.
* patient without sensory disorders
* patient with established organic of erectile dysfunction

Exclusion Criteria:

* investigator's impression of expected poor patient compliance or anatomic inadequacy (penile size/girth)
* Premature ejaculation
* Any psychiatric disorder
* Epilepsy
* Peyronie 's disease/ penile curvature
* Coagulopathy
* Any tumor in the pelvic or penile region within the last 3 years

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The OhhMed device provide treatments for improvement of erectile dysfunction
Enrollment: 28 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Change in erectile function (EF) | Baseline to 1 month post intervention
  The International Index for Erectile Function (IIEF) questionnaire will be administered. This is a 15 item tool; 6 ask questions addressing Erectile function over the previous 4 weeks. Scores from 0-30 can be obtained in this domain. Scores are interpreted as follows: 0-6 = Severe dysfunction, 7-12 = Moderate dysfunction, 13-18 = mild-moderate dysfunction, 19-24 = mild dysfunction, 25-30 = No dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Gruenwald, Prof., Principal Investigator — Rambam Medical Center, Haifa Israel
Locations (1):
- Rambam Medical center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No